CLINICAL TRIAL: NCT00924430
Title: A Drug Interaction Study to Investigate the Effects of SLV337 on the Pharmacokinetics of Simvastatin and Simvastatin Acid in Healthy Male Volunteers
Brief Title: Interaction Study SLV337/Simvastatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Responsible Party: Claire Nee, Solvay Pharmaceuticals
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S337.1.002; 2009-010392-24
Record Dates: First submitted 2009-05-19; First posted 2009-06-19 (Estimated); Last update posted 2009-09-09 (Estimated); Status verified 2009-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Interaction SLV337 and simvastatin; Type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other)
  Interventions: Drug: Simvastatin- SLV337 SD beta- SLV337 SD alpha - SLV337 MD beta- SLV337 SD beta+ Simvastatin
- 2 (Other)
  Interventions: Drug: Simvastatin - SLV337 SD alpha - SLV337 SD beta - SLV337 MD beta - SLV337 SD beta+ Simvastatin

INTERVENTIONS:
Drug: Simvastatin- SLV337 SD beta- SLV337 SD alpha - SLV337 MD beta- SLV337 SD beta+ Simvastatin — Single dose of 40 mg simvastatin tablet, single dose of 1400 mg SLV337 beta capsule, single dose of 1400 mg SLV337 alpha capsule, multiple dose over 12 days of 1400 mg/day SLV337 beta capsule including a single dose of 40 mg simvastatin tablet before the last dosing day
  Arms: 1
Drug: Simvastatin - SLV337 SD alpha - SLV337 SD beta - SLV337 MD beta - SLV337 SD beta+ Simvastatin — Single dose of 40 mg simvastatin tablet, single dose of 1400 mg SLV337 alpha capsule, single dose of 1400 mg SLV337 beta capsule, multiple dose over 12 days of 1400 mg/day SLV337 beta capsule including a single dose of 40 mg simvastatin tablet before the last dosing day
  Arms: 2

SUMMARY:
To investigate the effect of multiple doses of SLV337 on the pharmacokinetics of simvastatin and simvastatin acid when co-administered in healthy male subjects

ELIGIBILITY:
Inclusion Criteria:

* Volunteers with Body Mass Index 18.0-28.0 kg/m2

Exclusion Criteria:

* Clinically relevant medical history

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2009-06; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Simvastatin and simvastatin acid: Cmax, tmax, AUC0-t, AUC, lz, and t1/2, as well as CL/F and Vz/F for simvastatin only | 20 days

SECONDARY OUTCOMES:
SLV337 and its acylglucuronide metabolite: Cmax, tmax, AUC0-24, AUC0-t, CL/F (SLV337 only) on Days 1 and 13, as well as AUC, lz, t1/2 and Vz/F (SLV337 only) on Day 1 | 20 days
Safety and tolerability assessments including adverse events, clinical laboratory tests, electrocardiogram (ECG) and vital signs | During the duration of study participation

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (1):
- Site 1, London, United Kingdom